CLINICAL TRIAL: NCT05347264
Title: Comparative Effects of Gun Massager and Transverse Friction Massage on Pain and Disability in Patients With Plantar Fasciitis
Brief Title: Comparative Effects of Gun Massager and Transverse Friction Massage in Patients With Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0146 Amna
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Plantar Fascitis
Keywords: plantar fasciitis; foot and ankle disability index; numeric pain scale; deep friction massage; gun massager
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- massage gun (Experimental): 15 to 20 minutes along with hot pack.
  Interventions: Other: gun massager
- transverse friction massage (Experimental): 15 to 20 minutes along with hot pack.
  Interventions: Other: transverse friction massage

INTERVENTIONS:
Other: gun massager — 15 to 20 minutes along with hot pack.
  Arms: massage gun
Other: transverse friction massage — 15 to 20 minutes along with hot pack.
  Arms: transverse friction massage

SUMMARY:
to compare the effects of massage gun and transverse friction massage on management of pain and disability in patients with plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of morning heel pain with taking first step.
* Patients with limited range of motion and diagnosed with plantar fasciitis.
* Patients who are willing to participate.

Exclusion Criteria:

* Patient with heel fracture and surgeries will be excluded.
* Patient with sign of local and generalized infection or sepsis.
* Patient with foot deformities will be excluded

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Numeric pain scale | 4th week
  used as pain measurement tool to measure intensity of pain with 0 to 10 points. 0 Indicates no pain while 10 indicates severe pain
Foot and ankle disability index | 4th week
  Foot and ankle disability index is an area of explicit self-report of capacity with 2 components to evaluate disability identified with explicit conditions. The index was first portrayed in 1999 by Martin they survey impairments of everyday living

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Aftab Hospital Daska, Daska Kalan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rittu SB. A Comparative study on the Effectiveness of Myofascial Release and Deep Friction Massage in the Management of Foot Function and Flexibility among Chronic Plantar Fasciitis Patients: RVS College of Physiotherapy, Coimbatore; 2016.
- [Background] Kashif M, Albalwi A, Alharbi A, Iram H, Manzoor N. Comparison of subtalar mobilisation with conventional physiotherapy treatment for the management of plantar fasciitis. J Pak Med Assoc. 2021 Dec;71(12):2705-2709. doi: 10.47391/JPMA.1049. PMID 35150524
- [Background] Fraser JJ, Corbett R, Donner C, Hertel J. Does manual therapy improve pain and function in patients with plantar fasciitis? A systematic review. J Man Manip Ther. 2018 May;26(2):55-65. doi: 10.1080/10669817.2017.1322736. Epub 2017 May 3. PMID 29686479
- [Background] Lakhwani M, Phansopkar P. Efficacy of Percussive massage Versus Calf Stretching on Pain, Range of Motion, Muscle Strength and Functional Outcomes in Patients with Plantar Fasciitis-A Randomized Control Trial. 2021.
- [Background] Fraser JJ, Glaviano NR, Hertel J. Utilization of Physical Therapy Intervention Among Patients With Plantar Fasciitis in the United States. J Orthop Sports Phys Ther. 2017 Feb;47(2):49-55. doi: 10.2519/jospt.2017.6999. PMID 28142368
- [Background] Moshrif A, Elwan M, Daifullah OS. Deep friction massage versus local steroid injection for treatment of plantar fasciitis: a randomized controlled trial. Egyptian Rheumatology and Rehabilitation. 2020;47(1):1-5.
- [Background] Jones ER, Finley MA, Fruth SJ, McPoil TG. Instrument-Assisted Soft-Tissue Mobilization for the Management of Chronic Plantar Heel Pain: A Pilot Study. J Am Podiatr Med Assoc. 2019 May;109(3):193-200. doi: 10.7547/16-105. Epub 2019 Mar 27. PMID 30916579
- [Background] Yelverton C, Rama S, Zipfel B. Manual therapy interventions in the treatment of plantar fasciitis: A comparison of three approaches. Health SA. 2019 Sep 25;24:1244. doi: 10.4102/hsag.v24i0.1244. eCollection 2019. PMID 31934436